CLINICAL TRIAL: NCT05281133
Title: Effect Of Virtual Reality Glasses Used During Splint Application On Children's Pain And Anxiety Levels.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Çağla Kaya, Principal Investigator, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KBU-SBE-CK-01
Record Dates: First submitted 2022-03-02; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Pain, Acute; Anxiety Acute; Fractures, Bone
Keywords: Anxiety; child; fracture; nurse; pain; splint; virtual reality glasses
MeSH Terms: conditions — Acute Pain; Fractures, Bone; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: The study was carried out as a randomized controlled. In the study, two groups consisted of experimental group (n=40) and control group (n=40) were determined.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A total of 80 children assigned by randomization method (experimental group=40, control group= 40) were included in the sample group. The "Participant Information Form", the "Practice Registration Form", the "Wong Baker Pain Scale", the "State Anxiety Inventory for Children", the "After Splint Child's General Condition Evaluation Form", virtual reality glasses and pulse oximeter were used to collect data by outcomes assessor. Pain, anxiety and vital signs of the children in the experimental and control groups were recorded before, during and after the splint. The video chosen by the children in the experimental group was started 1-2 minutes before the splint with virtual reality glasses and watched for an average of 7 minutes. In the control group, during the splint a video was not watched.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group using virtual reality glasses (Experimental): The video chosen by the children in the experimental group was started 1-2 minutes before the splint with virtual reality glasses and watched for an average of 7 minutes.
  Interventions: Other: The group using virtual reality glasses
- The group not using virtual reality glasses (No Intervention): In the control group, during the splint a video was not watched.

INTERVENTIONS:
Other: The group using virtual reality glasses — The video chosen by the children in the experimental group was started 1-2 minutes before the splint with virtual reality glasses and watched for an average of 7 minutes.
  Arms: The group using virtual reality glasses

SUMMARY:
The study in order to evaluate the effect of virtual reality glasses during splint in children on pain and anxiety due to the procedure.

DETAILED DESCRIPTION:
The study was carried out as a randomized controlled experimental study in order to evaluate the effect of virtual reality glasses during splint in children aged 6-12 years on pain and anxiety due to the procedure.

The sample of the research consisted of 80 childrens who came to Karabuk University Training and Research Hospital orthopedic policlinic and emergency between 1 May and 31 October 2021 for the splint application. In the study, two groups consisted of experimental group (n=40) and control group (n=40) were determined.

The "Participant Information Form", the "Wong Baker Pain Scale", the "State Anxiety Inventory for Children", virtual reality glasses and pulse oximeter were used to collect data. The pain, anxiety and vital signs of the children in the experimental and control groups were recorded before, during and after the splint.

The video chosen by the children in the experimental group was shown with virtual reality glasses during the splint application. In the control group a video wasn't shown during the splint application. Chi square, Mann Whitney U, Bonferroni and Friedman tests were used in the analysis of data.

ELIGIBILITY:
Inclusion Criteria:

* The child should be between the ages of 6 and 12 age old.
* Acceptance of the research and giving written consent by the family and the child.
* Ability of the family and child to speak Turkish.
* The child should not wear glasses.
* The child should be at a cognitive level able to choose videos.

Exclusion Criteria:

* The child should have chronic diseases.
* The child should take analgesics with in the last 24 hours.
* The child should have physical, mental and neurological disabilities.
* The child has a febrile illness.
* Fainting of the child during the procedure.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Wong Baker Pain Scale- (FACES) | six months
  Wong Baker Faces Pain Rating Scale was developed by Wong and Baker (1981) and was reorganized in 1983. It is employed in the diagnosis of pain severity in 3e18 years-old children. It includes a zero (0) to five (5) scoring system. It is a horizontal scale of 6 hand-drawn faces, from 0 to 5, that range from a smiling "no hurt" face on the left followed by "hurts little bit", "hurts little more", "hurts even more", "hurts whole lot" to a crying "hurts worst" face on the right and scoring is conducted according to the image.
State-Trait Anxiety Inventory for Children- (STAI-CH) | six months
  State-Trait Anxiety Inventory for Children is the scale developed Spielberg's (1966) for testing anxiety. Children are asked to assess how they feel at the moment and to mark the most appropriate option. For each of the 20 items to evaluate the level of anxiety, one of the options (scored as 1, 2 or 3) is marked according to the presence and severity of the symptom. Turkish adaptation, validity and reliability study of this scale was done by Şeniz Özusta (1993). The scale, which consists of twenty items, aims to evaluate the emotions associated with state anxiety such as tension, nervousness, perturbation, and haste. When the presence of these emotions is reported as "very much so" by the child, the highest score is 3 and the lowest score of 1is assigned when "not at all" is preferred. The highest score in the scale is 60 and the lowest score is 20.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Öztürk Şahin, ass. prof., Study Director — Karabuk University
Locations (1):
- Institute of Health Sciences Karabuk University, Karabük, Merkez/Turkey, Turkey (Türkiye)